CLINICAL TRIAL: NCT00460993
Title: Efficacy and Safety of Eszopiclone (Lunesta) in Nursing Home Patients
Brief Title: Efficacy & Safety of Eszopiclone (Lunesta) in Nursing Home Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia C Griffiths, Principal Investigator, Emory University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 057-2006; LunestaNH (Other: Sepracor)
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Poor Quality Sleep
Keywords: Aging; Sleep; Nursing Home; Sleep in nursing homes
MeSH Terms: interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Lunesta Active drug (eszopiclone) 1 mg during 1st week of active drug. If sleep efficiency does not improve does increases to 2 mg for 2nd week of active drug administration.
  Interventions: Drug: Lunesta
- Group 2 (Placebo Comparator): Sugar pill packaged and supplied by Sepracor. One pill weeks one and two of intervention.
  Weeks 3 and 4 this Placebo group crosses over to active drug. 1 mg week 3 increasing to 2mg week 4 if sleep efficiency does not improve.
  Interventions: Drug: Lunesta

INTERVENTIONS:
Drug: Lunesta — Both groups receive eszopiclone. Group 1 receives Lunesta (eszopiclone) in intervention weeks 1 and 2 followed by placebo in weeks 3 and 4.
  Group 2 receives placebo in intervention weeks one and two followed by Lunesta (eszopiclone) in weeks 3 and 4.
  Other Names: eszopiclone

SUMMARY:
The purpose of this study is to examine the effects of the sleep aid Lunesta (Eszopiclone), on older adults who reside in a nursing home and have poor sleep as determined by wrist actigraphy.

DETAILED DESCRIPTION:
Older people living in nursing homes do not sleep very well for many reasons including pain, sleep disorders like sleep apnea (when someone briefly stops breathing during sleep) and night time urination, as well as the environmental disturbances caused by living in the nursing home, such as noise and disruptive care routines. Previous studies' attempts to improve sleep by modifying the nighttime nursing home environment have shown limited improvements in sleep.

This study will evaluate how well eszopiclone (Lunesta) works to improve sleep in nursing home residents with poor sleep. Eszopiclone is FDA approved and has been tested on older adults living in the community, but not on older adults living in nursing homes. We expect sleep to improve on the study drug, in comparison to the placebo. Based on adverse events reported in previous samples of older subjects, we expect the study drug to cause very few side effects.

We will evaluate how well eszopiclone works by measuring sleep at night and during the day. After consenting and final determination of eligibility, participants will complete a baseline phase to assess typical sleep, as well as daytime alertness and activity, thinking, memory and mood. Sleep at night and during the day will be objectively assessed with wrist actigraphs for all subjects. Approximately half will also receive polysomnographic studies to assess nighttime sleep. Subjects who sleep more than 75% of the time they are in bed will not continue in the study. Subjects will be randomized to one of two treatment groups-one will receive the active drug and then a placebo and the other will receive the placebo first and then the active drug. Following randomization, subjects will complete a brief run-in phase and then enter the treatment phase. Assessment of sleep and other measures will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Nursing Home Patients
* Age 65 and above

Exclusion Criteria:

* Under age 65
* Anticipated short stay (short term or hospice)
* Severe behavioral disturbance
* Unstable drug regimen in prior 2 weeks
* Use of a hypnotic, antihistamine, benzodiazepine, narcotic or antipsychotic

  * once per week in prior 2 weeks
* Use of a potent inhibitor of CYP3A4
* Parkinson's with uncontrolled tremor
* Severe Dementia
* Severe Sleep Apnea
* Inability to tolerate wrist Actigraphy
* Sleep Efficiency >75%
* Sleep apnea
* Sleep efficiency of greater than 75% during the night.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Griffiths, PhD., Principal Investigator — Emory University

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Active drug during phase 1, then placebo during phase 2. Lunesta Active drug (eszopiclone) 1 mg for 3 days. If sleep efficiency does not improve in 3 three day, dose increases to 2 mg for the next three days of active drug administration.
- Group 2: Placebo during phase 1, then active drug phase 2. One placebo for 6 days
Period: Phase 1 (6 Days)
Arm/Group | Group 1 | Group 2
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0
Period: Phase 2 (6 Days)
Arm/Group | Group 1 | Group 2
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 71 subjects were in baseline. But only 31 subjects enrolled into the study intervention portion used for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.1 (8.5) | 88.9 (5.6) | 86.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31
Sleep Efficiency [Median (Full Range); unit: percent of sleep] | 56.1 [28.2 to 74.9] | 60.7 [12.3 to 70.8] | 59.1 [12.3 to 74.9]

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency
Description: Percentage of time in bed at night asleep, averaged over 3 nights, as measured by actigraphy (and by polysomnography in a subgroup of subjects), holding constant time in bed and recording time
Time Frame: 6 days
Measure: Median (Full Range); unit: percentage of sleep
Groups:
- Group 1: Active drug given in phase 1, then Placebo pill in phase 2. Lunesta Active drug (eszopiclone) 1 mg during three days of active drug. If sleep efficiency does not improve doses increases to 2 mg for the next three days of active drug administration.
- Group 2: Placebo pill in phase 1, then Active drug given in phase 2. One placebo pill for 6 days
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 17
percentage of sleep | 70.0 [18.1 to 85.2] | 65.8 [16.0 to 83.5]

ADVERSE EVENTS:
Groups:
- Group 1: Active drug given in phase 1, then placebo pill given in phase 2.
- Group 2: Placebo pill given in phase 1, then active drug give in phase 2. One placebo pill for 6 days.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17

LIMITATIONS AND CAVEATS:
Low power to detect statistically significant effects of the interventions on outcomes; Inability to examine predictors of responsiveness because of the small sample size and the large number of predictors of response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No